CLINICAL TRIAL: NCT06647706
Title: Prevalence and Risk Factors of Pulmonary Hypertension in Patients with Myeloproliferative Neoplasms in Assiut University Hospital.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrhman Khalaf Hadyia Mohamed, dr, Assiut University
Other Study IDs: Prevalence of PH in MPNs
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Myeloproliferative Neoplasm
Keywords: pulmonary HTN; MPNs
MeSH Terms: conditions — Myeloproliferative Disorders | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MPNs patients who have echocardiographic probability of PH: MPNs patients who have echocardiographic probability of PH
  Interventions: Device: Transthoracic echocardiography
- MPNs patients who do not have echocardiographic probability of PH: MPNs patients who do not have echocardiographic probability of PH
  Interventions: Device: Transthoracic echocardiography

INTERVENTIONS:
Device: Transthoracic echocardiography — MPNs patients who have echocardiographic probability of PH

SUMMARY:
This study will evaluate the MPNs patients for the presence of PH by using a non invasive method ( Transthoracic echocardiography (TTE )) and correlate the clinical and laboratory data of these patients with development of PH aiming to identify risk factors for PH and parameters that can predict PH in MPNs patients and thus,identifying MPNs patients who require close monitoring & screening for PH ,hoping that early detection and management of PH in MPNs patients can improve morbidity, prognosis and survival in those patients.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a syndrome characterized by marked remodeling of the pulmonary vasculature and a progressive increase in the pulmonary vascular load. PH is a serious complex disorder that associated with high morbidity and mortality rates.

PH is a complication of various hematologic diseases including myeloproliferative neoplasms (MPNs) which are included in group 5 ph.

Myeloproliferative neoplasms (MPNs) are a group of diseases characterized by uncontrolled proliferation of at least one myeloid series due to an abnormal hematopoietic cell clone. There are different types of MPNs including polycythemia vera (PV), essential thrombocythemia (ET), chronic myeloid leukemia (CML), and primary myelofibrosis (PMF).

PH is defined as an elevation in the mean pulmonary artery pressure (mPAP) that is greater than or equal to 25 mmHg, which was measured at rest via right heart catheterization (RHC).

Systolic pulmonary artery pressure (sPAP) can be accurately estimated using Doppler transthoracic echocardiography (TTE), recent advances in noninvasive imaging led Doppler TTE to become the most widespread and well-recognized technique for non-invasive sPAP evaluation and the screening modality of choice for evaluating PH.

Active monitoring of PH in patients with MPN may be warranted. Identification of risk factors predicting PH in MPN patients promises early detection and possibly improved PH management and therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years)
2. patients diagnosed with MPNs. including polycythemia vera (PV), essential thrombocythemia (ET), chronic myeloid leukemia (CML), and primary myelofibrosis (PMF)

Exclusion Criteria:

1. patients less than 18 years old.
2. patients with cardiac diseases involving the left side of the heart or congenital heart diseases.
3. patients with chronic lung disease and primary pulmonary hypertension.
4. patients with chronic kidney disease.
5. patients with inherited and acquired chronic hemolytic anemia.
6. patients with connective tissue diseases.
7. patients with with past or current pulmonary embolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Assiut University Hospitals. (internal medicine Department and Outpatient Hematology Clinic )
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
determine the prevalence of pulmonary hypertension in patients with MPNs at Assiut University Hospital | 1 year
  To determine the prevalence of pulmonary hypertension in patients with MPNs at Assiut University Hospital by using a non invasive method ( Transthoracic echocardiography (TTE ))

SECONDARY OUTCOMES:
predictors of pulmonary hypertension in MPNs patients | 1 year
  To find the predictors of pulmonary hypertension through analysis of the data of those patients

REFERENCES:
- [Background] Humbert M, Kovacs G, Hoeper MM, Badagliacca R, Berger RMF, Brida M, Carlsen J, Coats AJS, Escribano-Subias P, Ferrari P, Ferreira DS, Ghofrani HA, Giannakoulas G, Kiely DG, Mayer E, Meszaros G, Nagavci B, Olsson KM, Pepke-Zaba J, Quint JK, Radegran G, Simonneau G, Sitbon O, Tonia T, Toshner M, Vachiery JL, Vonk Noordegraaf A, Delcroix M, Rosenkranz S; ESC/ERS Scientific Document Group. 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension. Eur Respir J. 2023 Jan 6;61(1):2200879. doi: 10.1183/13993003.00879-2022. Print 2023 Jan. No abstract available. PMID 36028254
- [Background] Ferrari A, Scandura J, Masciulli A, Krichevsky S, Gavazzi A, Barbui T. Prevalence and risk factors for Pulmonary Hypertension associated with chronic Myeloproliferative Neoplasms. Eur J Haematol. 2021 Feb;106(2):250-259. doi: 10.1111/ejh.13543. Epub 2020 Nov 22. PMID 33135220
- [Background] Lafitte S, Pillois X, Reant P, Picard F, Arsac F, Dijos M, Coste P, Dos Santos P, Roudaut R. Estimation of pulmonary pressures and diagnosis of pulmonary hypertension by Doppler echocardiography: a retrospective comparison of routine echocardiography and invasive hemodynamics. J Am Soc Echocardiogr. 2013 May;26(5):457-63. doi: 10.1016/j.echo.2013.02.002. Epub 2013 Mar 16. PMID 23510536
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Respir J. 2015 Oct;46(4):903-75. doi: 10.1183/13993003.01032-2015. Epub 2015 Aug 29. PMID 26318161
- [Background] Lahm T, Chakinala MM. World Health Organization group 5 pulmonary hypertension. Clin Chest Med. 2013 Dec;34(4):753-78. doi: 10.1016/j.ccm.2013.08.005. Epub 2013 Oct 18. PMID 24267303
- [Background] Simonneau G, Gatzoulis MA, Adatia I, Celermajer D, Denton C, Ghofrani A, Gomez Sanchez MA, Krishna Kumar R, Landzberg M, Machado RF, Olschewski H, Robbins IM, Souza R. Updated clinical classification of pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D34-41. doi: 10.1016/j.jacc.2013.10.029. PMID 24355639
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254